CLINICAL TRIAL: NCT01748526
Title: A Single-Dose, Open-Label, Randomized, Two-Way, Cross-Over Study to Assess the Pharmacokinetics and Pharmacodynamics of JNJ-28431754 in Healthy Indian Subjects
Brief Title: A Study to Assess the Pharmacokinetics and Pharmacodynamics of Canagliflozin (JNJ-28431754) in Healthy Indian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR014986; 28431754DIA1008 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Pharmacodynamics; Indian
MeSH Terms: interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Each volunteer will receive a single 200 mg dose of canagliflozin (JNJ-28431754) on Day 1.
  Interventions: Drug: Canagliflozin (JNJ-28431754) 200 mg
- Treatment B (Experimental): Each volunteer will receive a single 300 mg dose of canagliflozin (JNJ-28431754) on Day 1.
  Interventions: Drug: Canagliflozin (JNJ-28431754) 300 mg

INTERVENTIONS:
Drug: Canagliflozin (JNJ-28431754) 200 mg — One 200 mg tablet taken orally (by mouth) on Day 1.
  Other Names: JNJ-28431754
  Arms: Treatment A
Drug: Canagliflozin (JNJ-28431754) 300 mg — One 300 mg tablet taken orally (by mouth) on Day 1.
  Other Names: JNJ-28431754
  Arms: Treatment B

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (ie, how the body affects the drug) and pharmacodynamics (ie, how the drug affects the body) of 2 different doses of canagliflozin (JNJ-28431754) in healthy Indian volunteers.

DETAILED DESCRIPTION:
This study will be an open-label (all volunteers and study staff know the identity of the assigned treatment), randomized (the treatment is assigned by chance), single center, single dose, 2-way cross-over study (all volunteers switch from one treatment to another) to assess the pharmacokinetics and pharmacodynamics of canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus) in healthy Indian volunteers. The study will consist of 3 phases: a single screening phase, a baseline phase of 2 days per period, and an open-label treatment phase that includes 2 treatment periods (Periods 1 and 2). During Period 1, volunteers will be randomly assigned to receive a single dose of either 200 mg (Treatment A) or 300 mg (Treatment B) of canagliflozin on Day 1. During Period 2, volunteers will receive the dose of canagliflozin (Treatment A or B) that they did not receive during Period 1. The duration of each treatment period will be 4 days and each treatment period will be separated by a 14 day washout period (when no medication is given). Each volunteer will participate in the study for approximately 45 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a body mass index (BMI = weight in kg/height in m2) between 18 and 35 kg/m2 (inclusive) and body weight not less than 50 kg
* Volunteer must have a glomerular filtration rate (the volume of fluid filtered by the kidney) more than or equal to 90 mL/min/1.73 m2 using the Modification of Diet in Renal Disease calculation
* Fasting blood glucose at screening must be less than 100 mg/dL and the 2 hour plasma glucose following the oral glucose tolerance test (conducted at screening) must be less than 140 mg/dL

Exclusion Criteria:

* History of or currently active illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results
* Female volunteer is breast-feeding
* Volunteer has a history of smoking or use of nicotine-containing substances within the previous 2 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin JNJ-28431754) | Up to Day 4
  Plasma concentrations of canagliflozin (JNJ-28431754), following the administration of a single 200mg dose and a single 300 mg dose, will be used to determine pharmacokinetic parameters for canagliflozin (measurements describing how the body affects the drug).
Urine concentrations of canagliflozin (JNJ-28431754) | Up to Day 4
  Urine concentrations of canagliflozin (JNJ-28431754), following the administration of a single 200mg dose and a single 300 mg dose, will be used to determine pharmacokinetic parameters for canagliflozin (measurements describing how the body affects the drug).
Change from baseline in 24-hour urine glucose excretion | Day -1 (Baseline) up to Day 3
  Change from baseline in 24-hour urine glucose excretion following the administration of a single 200 mg dose and a single 300 mg dose of canagliflozin (JNJ-28431754) will be used to evaluate the pharmacodynamics of canagliflozin (ie, how the drug affects the body).
Change from baseline in the area under the plasma glucose concentration-time curve (AUC) | Day -1 (Baseline) and 4 hours post-dose
  Change from baseline in the area under the plasma glucose concentration-time curve (AUC) (a measure of the body's exposure to glucose) at 4 hours following the administration of a single 200mg dose and a single 300 mg dose of canagliflozin (JNJ-28431754) will be used to assess the pharmacodynamics of canagliflozin (ie, how the drug affects the body).
Change from baseline in the area under the plasma insulin concentration-time curve (AUC) | Day -1 (Baseline) and 4 hours post-dose
  Change from baseline in the area under the plasma insulin concentration-time curve (AUC) (a measure of the body's exposure to insulin) at 4 hours following the administration of a single 200mg dose and a single 300 mg dose of canagliflozin (JNJ-28431754) will be used to assess the pharmacodynamics of canagliflozin (ie, how the drug affects the body).
Change from baseline in the area under the plasma C-peptide concentration-time curve (AUC) | Day -1 (Baseline) and 4 hours post-dose
  Change from baseline in the area under the plasma C-peptide concentration-time curve (AUC) (a measure of the body's exposure to C-peptide) at 4 hours following the administration of a single 200mg dose and a single 300 mg dose of canagliflozin (JNJ-28431754) will be used to assess the pharmacodynamics of canagliflozin (ie, how the drug affects the body).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Ahmedabad, India

REFERENCES:
- [Derived] Devineni D, Polidori D, Curtin C, Stieltjes H, Tian H, Wajs E. Single-dose Pharmacokinetics and Pharmacodynamics of Canagliflozin, a Selective Inhibitor of Sodium Glucose Cotransporter 2, in Healthy Indian Participants. Clin Ther. 2016 Jan 1;38(1):89-98.e1. doi: 10.1016/j.clinthera.2015.11.008. Epub 2015 Dec 11. PMID 26687552
- See also: A Single-Dose, Open-Label, Randomized, Two-Way, Cross-Over Study to Assess the Pharmacokinetics and Pharmacodynamics of JNJ-28431754 in Healthy Indian Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=2204&filename=CR014986_CSR.pdf